CLINICAL TRIAL: NCT05060601
Title: Healing of Periodontal Pockets Following Treatment With Minimally Non Surgical Approach or Conventional Non Surgical Therapy. A Randomized Controlled Clinical Trial
Brief Title: Minimally Non Surgical Periodontal Therapy Compared to Traditional Approach
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Luca Ramaglia, Professor Luca Ramaglia, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 465/20
Record Dates: First submitted 2021-09-06; First posted 2021-09-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Periodontal Diseases; Periodontal Inflammation
Keywords: Periodontitis; Osseous defects; Periodontal therapy
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gracey micro-curettes (Experimental): Subgingival mechanical debridement will be performed using an ultrasonic scaler with specific thin tips and Gracey micro-curette.
  Interventions: Procedure: Gracey micro-curettes
- Standard Gracey curettes (Active Comparator): Subgingival mechanical debridement will be performed using a conventional ultrasonic scaler and standard Gracey curettes.
  Interventions: Procedure: Standard Gracey curettes

INTERVENTIONS:
Procedure: Gracey micro-curettes — Mechanical debridement will be performed by means of ultrasonic scalers with specific thin tips and micro-curettes, in order to minimize trauma for gingival tissues.
  Arms: Gracey micro-curettes
Procedure: Standard Gracey curettes — After local anaesthesia, non surgical subgingival debridement will be performed by standard Gracey curettes
  Arms: Standard Gracey curettes

SUMMARY:
This study aims to evaluate the clinical results of non-surgical periodontal therapy performed with micro-instruments compared to traditional approach (standard curettes) after 6 months of follow-up.

The patients enrolled, subject to written informed consent, will be divided into a Test group (T) and a Control group (C) through a randomization process. Both groups will be motivated on the rules of oral hygiene, treated scrupulously and monitored monthly for 6 months, at the end of which the final data will be collected for statistical processing (in particular by analyzing the difference between baseline and after 6 months of the parameter "probing depth" or PD).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the clinical results of non-surgical periodontal therapy performed with micro-instruments (micro-curettes) compared to traditional instruments (standard curettes) after 6 months of follow-up.

The proposed clinical trial will be conducted according to the principles of the Declaration of Helsinki on experimentation involving human subjects.

All subjects will be recruited from the Area of Odontostomatology - Department of Neuroscience, Reproductive and Odontostomatological Sciences of the University of Naples "Federico II".

In a first phase, all patients will be treated with a supragingival scaling session in order to remove plaque and tartar and it will be provided instructions for a correct oral hygiene. After 1 week, the clinical parameters (PD, FMPS, FMBS, CAL, REC) will be recorded and the subjects randomly assigned to the Test (T) or Control (C) group.

In the Test group, after local anesthesia, subgingival mechanical debridement will be performed using an ultrasonic scaler with specific thin tips and Gracey micro-curette to minimize soft tissue trauma.

In the Control group, after local anesthesia, debridement will be performed using an ultrasonic scaler with specific thin tips and standard Gracey curettes.

At the end of the periodontal therapy, a polishing paste will be applied supragingival in both groups using a rubber cup. An antiseptic therapy based on mouthwash with chlorhexidine digluconate 0.12% (two rinses a day for the first two weeks) will then be recommended. No antibiotics will be prescribed.

Patients from both groups will be called up every month for a professional supragingival cleaning and professional motivation. The final evaluation will be carried out 6 months after the subgingival treatment.

Data analysis will be performed using statistical software (NCSS-PASS, NCSS, Kaysville, UT). The patient will be considered as a statistical unit; however an additional analysis based on the specific dental site will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Untreated patients diagnosed with severe/advanced periodontitis with slow/moderate rate of progression
* Age > 18 years
* Patients at least 10 teeth per arch
* Presence at least of two teeth with PD > 5 mm per quadrant
* Single-rooted teeth or multi-rooted without furcation involvement

Exclusion Criteria:

* Patients with systemic diseases
* Pregnant or lactating
* Tobacco smokers (<10 cigarettes/day)
* Previous periodontal treatment in the last 2 years
* Prolonged antibiotic treatment or anti-inflammatory treatment within 6 months prior to periodontal therapy
* Furcation involvement
* Acute periodontal or endodontic abscesses
* Third molars

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Change of Probing Depth (PD) (millimeters) | baseline, 1 week after supragingival scaling, 6 months after non-surgical periodontal therapy
  The distance from gingival margin to the bottom of the pocket

SECONDARY OUTCOMES:
Change of Full-Mouth Plaque Score (FMPS) (percentage) | baseline, 1 week after supragingival scaling, 6 months after non-surgical periodontal therapy
  Percentage of tooth sites revealing the presence of plaque
Change of Full-Mouth Bleeding Score (FMBS) (percentage) | baseline, 1 week after supragingival scaling, 6 months after non-surgical periodontal therapy
  Percentage of tooth sites revealing the presence of bleeding on probing
Change of Clinical Attachment Level (CAL) (millimeters) | baseline, 1 week after supragingival scaling, 6 months after non-surgical periodontal therapy
  Distance from the cement-enamel junction to the bottom of the pocket and gingival recession
Change of Gingival Recession (GR) (millimeters) | baseline, 1 week after supragingival scaling, 6 months after non-surgical periodontal therapy
  Distance from gingival margin to the cement-enamel junction

IPD SHARING:
Plan to Share IPD: No